CLINICAL TRIAL: NCT04783038
Title: The Effect of Distance Reiki on Patient Reported Quality of Life, Correlated With Changes in Immune Repertoires Among Multiple Myeloma Patients: A Pilot Study
Brief Title: Determining The Impact Of Distance Reiki On Patient Reported QOL And Immunity Among Multiple Myeloma Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 20-007168; NCI-2021-13433 (Registry Identifier: CTRP (Clinical Trials Reporting Program))
Record Dates: First submitted 2021-01-28; First posted 2021-03-04 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Multiple Myeloma; Autologous Stem Cell Transplant
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Who Masked: Investigator
Masking Description: This is a single blinded randomization to True Reiki therapy, Sham reiki Therapy or No intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Distance Reiki (Active Comparator): Subjects will be scheduled for once a week session of distance Reiki for 4 weeks.
  Interventions: Other: Distance Reiki
- Sham Reiki (Sham Comparator): Subjects will be scheduled for once a week session of Sham distance Reiki for 4 weeks.
  Interventions: Other: Sham distance Reiki
- Standard of Care (No Intervention): Subjects will not receive any Reiki treatment

INTERVENTIONS:
Other: Distance Reiki — Reiki therapy session performed remotely over a Zoom® video conferencing platform led by Reiki Practitioners who are also Health Care Providers at the Mayo Clinic, and have at least 6 months of experience in Reiki.
  Arms: Distance Reiki
Other: Sham distance Reiki — Session performed remotely over a Zoom® video conferencing platform led by a Health Care Provider employed at the Mayo Clinic, but will have no experience in Reiki and will not be a certified Reiki Practitioner.
  Arms: Sham Reiki

SUMMARY:
This research study is being done to determine if Distance Reiki therapy offers a quality of life benefit, and improves immunity compared to patients receiving Sham Distance Reiki therapy or no additional Reiki intervention.

DETAILED DESCRIPTION:
Reiki is a popular complementary medicine modality sought after by patients. This non- intrusive Japanese based therapy centers on the guiding of energy through a Reiki practitioner to the patient which facilitates innate healing by modulation of energy fields. Reiki is formally classified as biofield therapy by the National Center for Complementary and Alternative Medicine (NCCAM).

Current research indicates that Reiki shows promise as a noninvasive healing tool for mind and body, particularly among patients with cancer. However, the data validating the effectiveness of Reiki integrated within a structured medical paradigm and the effect on cancer immunity remains unknown.

Given the clear demand for Reiki among cancer patients but skepticism within the medical community, this trial will aim to determine an objective patient reported quality of life (PRQoL) benefit by utilizing validated tools, in order to effectively implement Reiki into traditional medical practice.

Multiple myeloma patients are at high risk of serious illness from the COVID-19 virus during this pandemic, and so distance Reiki will be carried out via video conferencing platform.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients with Multiple Myeloma with stable disease or currently in maintenance therapy
* English Speaking
* Computer and internet access with video conferencing availability

Exclusion Criteria:

* Evidence of disease relapse at the post-transplant follow up visit
* Patient not returning to Mayo Clinic Rochester for subsequent post-transplant follow up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-01-27 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Change in patient-reported quality of life | Baseline, approximately 5 weeks
  Measured using the Patient-Reported Outcomes Measurement Information System (PROMIS)-29 survey. PROMIS measures are scored on the T-score metric. High scores mean more of the concept being measured (eg. more Fatigue, more Physical Function)
Change in patient-reported overall quality of life | Baseline, approximately 5 weeks
  Measured using the single item Linear Analogue Self-Assessment (LASA) that uses a 10-point Likert scale, where 0=as bad as it can be and 10=as good as it can be
Acceptability of Distance Reiki among multiple myeloma (MM) outpatients. | Approximately 5 weeks
  Measured by using the "Was it worth it" (WIWI) questionnaire which patients will complete upon study completion. This is a 3 item questionnaire which assesses patient satisfaction. Higher scores indicate greater acceptability of the Reiki intervention.

SECONDARY OUTCOMES:
Phenotypic characterization of circulating immune cells | Baseline, approximately 5 weeks
  Measured using mass cytometry by time of flight (CyTOF) to phenotypically characterize the immune cells in peripheral blood
Assessment of T-cell receptor repertoire and T-cell clonal diversity | Baseline, approximately 5 weeks
  Analyzed using multiplex polymerase chain reaction (PCR) RNA-sequencing to define T-cell antigen receptor (TCR) repertoire.

CONTACTS AND LOCATIONS:
Overall Officials: Martha Lacy, MD, Principal Investigator — Mayo Clinic; Joselle M. Cook, MBBS, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials